CLINICAL TRIAL: NCT03488316
Title: Influence of Temporary Filling Material Composition on the Success Rate of Endodontic Treatments - Randomized Clinical Study
Brief Title: Influence of Temporary Filling Material Composition on the Success Rate of Endodontic Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PAULO VINICIUS SOARES (Other)
Responsible Party: Sponsor-Investigator, PAULO VINICIUS SOARES, Director of NCCL Research Group, Federal University of Uberlandia
Organization: Federal University of Uberlandia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.527.632
Record Dates: First submitted 2018-03-06; First posted 2018-04-05 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: MTA; Calcium Hydroxide; Endodontic Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide temporary filling material (Active Comparator): Temporary filling with Ca(OH)2
  Interventions: Procedure: Carie removal; Procedure: Absolute isolation; Drug: Manipulation of the temporary filling material based on Calcium Hydroxide; Procedure: Material insertion on the root canal; Procedure: Material re-insertion on the root canal accordging to the infection needs.; Procedure: Definiteve canal root obturation; Procedure: Definitve restoration
- MTA temporary filling material (Active Comparator): Temporary filling with MTA
  Interventions: Procedure: Carie removal; Procedure: Absolute isolation; Drug: Manipulation of the temporary filling material based on Mineral trioxide aggregate; Procedure: Material insertion on the root canal; Procedure: Material re-insertion on the root canal accordging to the infection needs.; Procedure: Definiteve canal root obturation; Procedure: Definitve restoration

INTERVENTIONS:
Procedure: Carie removal — Carie removal with a low speed handpiece
Procedure: Absolute isolation — Absolute isolation with rubber dam
Drug: Manipulation of the temporary filling material based on Calcium Hydroxide — Manipulation of the temporary material based on Calcium Hydroxide according to the manufacturer's recommendations.
  Arms: Calcium Hydroxide temporary filling material
Drug: Manipulation of the temporary filling material based on Mineral trioxide aggregate — Manipulation of the temporary material based on Mineral trioxide aggregate according to the manufacturer's recommendations.
  Arms: MTA temporary filling material
Procedure: Material insertion on the root canal — Material insertion on the root canal according to the manufacturer's recommendations
Procedure: Material re-insertion on the root canal accordging to the infection needs. — Material re-insertion on the root canal according to the manufacturer's recommendations
Procedure: Definiteve canal root obturation — Definiteve canal root obturation with gutta-percha and definitive cement.
Procedure: Definitve restoration — Definitve restoration confecction.

SUMMARY:
The aim of this study is through a randomized clinical trial, double blind, splitmouth, evaluate the success rate (contamination rate, periapical lesion relapse and the presence of exudate between the treatment's sessions) of endodontically treated teeth that required filling with temporary material. The composition of the temporary filling material (cement (Based on calcium hydroxide; and based on mineral trioxide aggregate) will be evaluated. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
The need for endodontic treatment is still very common in the clinical routine, whether due to dento-alveolar trauma or caries. In some cases, the temporary filling procedure is required until the endodontic treatment is completed. The temporary filling material should be biocompatible and bacteriostatic. The aim of this study is through a randomized clinical trial, double blind, split-mouth, evaluate the success rate (contamination rate, periapical lesion relapse and the presence of exudate between the treatment's sessions) of endodontically treated teeth that required filling with temporary material. The composition of the temporary filling material (cement (Based on calcium hydroxide; and based on mineral trioxide aggregate) will be evaluated. Twenty participants with at least two teeth with the need of endodontic treatment will be selected. The teeth will be randomly divided into 2 different groups according to the temporary filling material composition (Based on calcium hydroxide; and based on mineral trioxide aggregate). Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Both genres
* Presence of at least two teeth with indication of endodontic treatment
* Good oral hygiene

Exclusion Criteria:

* Dentures or orthodontics
* Presence of periodontal disease
* Presence of parafunctional habits
* Presence of systemic disease
* Presence of severe psychological disturbe;
* Constant use of analgesic and, or anti-inflammatory
* Allergic response to dental products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Contamination rate of endodontically treated teeth that required filling with temporary material with a 1 year follow up. | 1 year
Periapical lesion relapse of endodontically treated teeth that required filling with temporary material with a 1 year follow up. | 1 year
Presence of exudate between the treatment's sessions of endodontically treated teeth that required filling with temporary material with a 1 year follow up. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett F. The role of endodontics in the treatment of luxated permanent teeth. Dent Traumatol. 2002 Apr;18(2):47-56. doi: 10.1034/j.1600-9657.2002.00098.x. PMID 12184211
- [Background] Camilleri J, Montesin FE, Brady K, Sweeney R, Curtis RV, Ford TR. The constitution of mineral trioxide aggregate. Dent Mater. 2005 Apr;21(4):297-303. doi: 10.1016/j.dental.2004.05.010. PMID 15766576
- [Background] da Rosa WLO, Cocco AR, Silva TMD, Mesquita LC, Galarca AD, Silva AFD, Piva E. Current trends and future perspectives of dental pulp capping materials: A systematic review. J Biomed Mater Res B Appl Biomater. 2018 Apr;106(3):1358-1368. doi: 10.1002/jbm.b.33934. Epub 2017 May 31. PMID 28561919
- [Background] Le Goff A, Bunetel L, Mouton C, Bonnaure-Mallet M. Evaluation of root canal bacteria and their antimicrobial susceptibility in teeth with necrotic pulp. Oral Microbiol Immunol. 1997 Oct;12(5):318-22. doi: 10.1111/j.1399-302x.1997.tb00397.x. PMID 9467386
- [Background] Malkoc MA, DemIr N, Sengun A, Bozkurt SB, Hakki SS. Cytotoxicity of temporary cements on bovine dental pulp-derived cells (bDPCs) using realtime cell analysis. J Adv Prosthodont. 2015 Feb;7(1):21-6. doi: 10.4047/jap.2015.7.1.21. Epub 2015 Feb 17. PMID 25722833
- [Background] Siqueira JF Jr, Rocas IN, Santos SR, Lima KC, Magalhaes FA, de Uzeda M. Efficacy of instrumentation techniques and irrigation regimens in reducing the bacterial population within root canals. J Endod. 2002 Mar;28(3):181-4. doi: 10.1097/00004770-200203000-00009. PMID 12017176
- [Background] Sjogren U, Figdor D, Persson S, Sundqvist G. Influence of infection at the time of root filling on the outcome of endodontic treatment of teeth with apical periodontitis. Int Endod J. 1997 Sep;30(5):297-306. doi: 10.1046/j.1365-2591.1997.00092.x. PMID 9477818
- [Background] Sundqvist G. Taxonomy, ecology, and pathogenicity of the root canal flora. Oral Surg Oral Med Oral Pathol. 1994 Oct;78(4):522-30. doi: 10.1016/0030-4220(94)90047-7. PMID 7800383
- [Background] von Arx T. [Mineral trioxide aggregate (MTA) a success story in apical surgery]. Swiss Dent J. 2016;126(6):573-95. doi: 10.61872/sdj-2016-06-02. French, German. PMID 27377433